CLINICAL TRIAL: NCT04744636
Title: Target Involvement and Exploratory Biomarkers Investigations in Healthy Volunteers and in Patients With Type 2 Diabetes Mellitus
Brief Title: Vascular Function and Biomarker Assessments in Healthy Volunteers and in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CL1-RTCMP-001; 2017-000045-42 (EudraCT Number)
Record Dates: First submitted 2021-01-27; First posted 2021-02-09 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Phase 1; Healthy volunteers; Clinical translational exploratory study; Target involvement; Exploratory biomarkers; Cardiovascular disease; Vascular function; Coronary flow reserve; Biopterins; Cutaneous blood flow
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy volunteers aged of 18-30 years (Other)
  Interventions: Drug: Other
- Healthy volunteers aged of 50-59 years (Other)
  Interventions: Drug: Other
- Healthy volunteers aged of 60-70 years (Other)
  Interventions: Drug: Other
- Type 2 diabetic patients aged of 50-70 years (Other)
  Interventions: Drug: Other

INTERVENTIONS:
Drug: Other — Healthy volunteers will be selected within 3 weeks before inclusion (Day 0). The investigations will be performed on 2 days (Day 1 (D1) and Day 2 (D2)): vascular endothelial function assessment and blood collection for biomarker investigation on Day 1 and Case Report Form (CFR) on Day 2.
  Then, subjects will be discharged at the end of the last investigation day (Day 2).
  All the participants have received two pharmacological agents (NIMP) :
  * Acetylcholine : administered subcutaneously (by iontophoresis) to assess maximal vascular endothelial function.
  * Adenosine : administered intravenously during MRI for the measurement of CFR.
  Arms: Healthy volunteers aged of 18-30 years; Healthy volunteers aged of 50-59 years; Healthy volunteers aged of 60-70 years
Drug: Other — Type 2 diabetic patients will be selected within 3 weeks before inclusion (Day 0).
  The investigations will be performed on 2 days (Day 1 (D1) and Day 2 (D2)): vascular endothelial function assessment and blood collection for biomarker investigation on Day 1 and CFR on Day 2.
  Then, subjects will be discharged at the end of the last investigation day (Day 2).
  All the participants have received two pharmacological agents (NIMP):
  * Acetylcholine : administered subcutaneously (by iontophoresis) to assess maximal vascular endothelial function.
  * Adenosine : administered intravenously during MRI for the measurement of CFR.
  Arms: Type 2 diabetic patients aged of 50-70 years

SUMMARY:
The purpose of this study is to evaluate the vascular function and biomarkers in healthy volunteers and type 2 diabetic patients.

DETAILED DESCRIPTION:
The present interventional study will be performed in 3 groups of healthy volunteers of different ages and in type 2 diabetic patients without an investigational medicinal product administrated.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Age [18 -30], [50-59] and [60-70] years
* Male and female healthy volunteers, except with skin types 5 and 6
* Body weight ≥ 50 kg and BMI between [18.0 -28.0] kg/m^2 inclusive
* Non or ex-smokers (defined as someone who completely stopped smoking for at least 1 month before the beginning of this study)
* No clinically relevant findings in the medical history and physical examination, especially with regards to cardiovascular system, lung, liver and renal function
* Normal blood and urine laboratory tests

Patients with type 2 diabetes (T2D) mellitus:

* Male and female patients, except with skin types 5 and 6
* Age [50 - 70] years
* BMI ≤35 kg/m2
* T2D patients (according to American Diabetes Association (ADA) criteria i.e. HbA1c > 6.5% or fasting plasma glucose > 126 mg/dL (7.00 mmol/L) or 2-hour glucose ≥ 200mg/dL (11.1mmol/L) after 75g oral glucose or glucose ≥200mg/dL (11.1mmol/L) at any time on two separate occasions (historic values and/or at selection)
* Currently treated with Standards of Medical Care in T2D at stable doses for at least 3 months
* Antihypertensive drugs allowed except beta-blockers and calcium antagonists
* Non or ex-smokers (defined as someone who completely stopped smoking for at least 1 month before the beginning of this study)

Non inclusion Criteria:

Healthy volunteers:

* Unlikely to co-operate in the study,
* Participation in another interventional study, including last study drug intake, at the same time or within the 3 months preceding the selection visit; participation in non-interventional registries or epidemiological studies is allowed,
* Deprived of his freedom by administrative or court order or under guardianship,
* History or evidence of acute or chronic abuse of alcohol consumption of> 21 alcohol units per week for males and >14 units per week for females (1 alcohol unit = 100 mL of 12% wine; = 30 mL of 40% spirits; = 250 mL of 6% beer),
* Positive alcohol breath test,
* Positive cotinine test,
* Known or suspected to be drug-dependent,
* Positive result in urinary screening for drug abuse,
* Pregnancy, breastfeeding or lactating,
* Regular use of prescribed and non-prescribed drugs in the last 60 days before the day of investigations into the study except hormonal contraception (e.g. pill or hormonal intrauterine device (IUD) or hormonal implants or Nuva Ring) (if applicable),
* Any drug intake of prescribed or non-prescribed drugs including over-counter drugs (except acetaminophen), herbal remedies or nutritional supplements such as multivitamins in the 2 weeks before the day of investigations unless the investigator deems this drug intake to be irrelevant for the purpose of this study and that can be temporarily suspended,
* Intake of dipyridamol (contraindicated with adenosine infusion)
* Known hypersensitivity to adenosine injection,
* Any acute or chronic illness or clinically relevant findings (i.e. liver, kidney, cardiovascular diseases) in the selection visit examinations,

Patients with type II diabetes mellitus (T2D):

* Unlikely to co-operate in the study,
* Participation in another interventional study, including last study drug intake, at the same time or within the 3 months preceding the selection visit; participation in non-interventional registries or epidemiological studies is allowed,
* Deprived of his freedom by administrative or court order or under guardianship,
* Unwilling to allow his or her primary care practitioner to be notified of participation in the study and for information on a participant's medical history to be obtained from the general practitioner,
* History or evidence of acute or chronic abuse of alcohol consumption of> 21 alcohol units per week for males and >14 units per week for females (1 alcohol unit = 100 mL of 12% wine; = 30 mL of 40% spirits; = 250 mL of 6% beer),
* Positive alcohol breath test,
* Positive cotinine test,
* Known or suspected to be drug-dependent,
* Positive result in urinary screening for drug abuse,
* Pregnancy, breastfeeding or lactating,
* Intake of dipyridamol (contraindicated with adenosine infusion)
* Known hypersensitivity to adenosine injection,
* Any acute or chronic illness or clinically relevant findings (i.e. liver,kidney, cardiovascular diseases) in the selection visit examinations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Guanylate triphosphate cyclohydrolase (GTP-CH) investigations | Day 1
  Plasma/platelet levels of Dihydrobiopterin (BAH)/Tetrahydrobiopterin (BH4), Cyclic guanosine monophosphate (cGMP)
Guanylate triphosphate cyclohydrolase (GTP-CH) investigations | Day 1
  Blood flow changes for vascular endothelial function
Guanylate triphosphate cyclohydrolase (GTP-CH) investigations | Day 2
  Coronary flow reserve
Guanylate triphosphate cyclohydrolase (GTP-CH) investigations | Day 1
  Genomic market (blood) DNA and/or RNA characteristics of genes such as GTP Cyclohydrolase 1 (GCH)

SECONDARY OUTCOMES:
Adverse events | Through study completion, 3.5 weeks
  Occurence of any adverse events
Blood pressure supine | Day 1
  Relevant abnormalities on supine blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Denis Strugala, Dr, Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/